CLINICAL TRIAL: NCT00971074
Title: The Use of Viscosupplementation for the Treatment of Patients With Persistent Non-mechanical Pain Status-post Partial Menisectomy
Brief Title: Study of Viscosupplementation for the Treatment of Knee Pain After Menisectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients did not meet inclusion criteria.
Sponsor: Grant Jones (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor-Investigator, Grant Jones, Associate Professor-Clinical, Orthopaedics, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009H0156
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Arthralgia
Keywords: Arthralgia; Viscosupplementation; Knee; Menisci, Tibial; Surgery, Outpatient
MeSH Terms: conditions — Arthralgia | interventions — hylan; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hylan G-F 20 (Experimental): Single injection of Hylan G-F 20 into the affected knee.
  Interventions: Drug: Hylan G-F 20
- Sham Injection (Sham Comparator): A needle will be inserted through the knee capsule but no medication will be injected.
  Interventions: Other: Sham Injection

INTERVENTIONS:
Drug: Hylan G-F 20 — 6 ml intra-articular injection given once. The injection takes approximately 15 seconds.
  Other Names: Synvisc One
  Arms: Hylan G-F 20
Other: Sham Injection — A needle will be inserted through the knee capsule but no medication will be injected.
  Arms: Sham Injection

SUMMARY:
The investigators' objective is to analyze a group of patients who have had a partial meniscectomy but continue to have knee pain after surgery with a double-blind, randomized prospective study comparing the use of Hylan G-F 20(single injection of a viscosupplementation) versus placebo injection. The investigators would expect patients who receive the treatment (Hylan G-F 20) to have lower pain compared to the patients who were in the placebo group (had the needle injected into the knee but no medication or substance injected) since Hylan G-F 20 has been shown to decrease pain in arthritic patients.

DETAILED DESCRIPTION:
A great majority of patients who have a partial menisectomy for mechanical symptoms do well with full return of function without pain. There is a sub-group of patients who are found to have Grade II- III chondromalacia lesions (deemed arthritic) at the time of surgery that have persistent generalized "arthritic-type" pain despite relief of their mechanical symptoms. To date, there are no published studies analyzing if this treatment is better than no treatment in this group of patients. We would expect patients who receive the treatment (Hylan G-F 20) to have lower pain compared to the patients who were in the placebo group (had the needle injected into the knee but no medication or substance injected) since Hylan G-F 20 has been shown to decrease pain in arthritic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* S/P partial medial and/or lateral partial meniscectomy
* Pre-operative MRI diagnosed meniscal tear
* Diffuse, non-focal arthroscopically diagnosed ICRS Grade II or III chondromalacia. (used to determine the presence of tibiofemoral osteoarthritis)
* Baseline VAS pain score between 50 and 80mm.
* Persistent, generalized knee pain without mechanical symptoms
* Kellgren/Lawrence (K/L) grade II or III (used to determine the presence of tibiofemoral osteoarthritis)

Exclusion Criteria:

* Bilateral arthroscopy (within 6 months pre- and post- initial VAS score.
* Complete meniscectomy
* Microfracture (via drilling, picking, abrading, thermal or radiofrequency or any procedure that violates the subchondral plate)
* Focal chondral lesion visualized on arthroscopy or any focal cartilage procedure (e.g. ACI, OATS, mosaicplasty, etc)
* Concomitant ligamentous injury or repair
* K/L stage I or IV
* Significant Varus or Valgus clinical malalignment
* S/P tibial osteotomy in target knee
* Isolated patello-femoral OA or isolated anterior knee pain
* Prosthetic implant in either knee
* Re-injury in time between original surgery and baseline visit
* Inflammatory arthritis (e.g. rheumatoid arthritis, gout, pseudogout (chondrocalcinosis), lupus, etc)
* Obesity with BMI > 35 (at time of initial VAS score
* NSAIDs or opiates within one week of baseline randomization or during trial period
* Known allergy to viscosupplements, known allergy to avian, egg or feather products
* Prior Viscosupplementation use in ipsilateral knee
* Oral steroids (within 4 weeks of initial VAS score)
* IA steroids in target knee within 6 months
* Significant medical co-morbidities ( e.g. malignancy, hepatic, renal, cardiac, pulmonary, gastrointestinal disease) in the judgment of the investigator
* Known hip disease
* Pregnant or nursing (at time of injection, pregnancy test at visit)
* Active infection of either lower extremity or past history of septic arthritis
* Venous or lymphatic stasis in either lower extremity
* Enrolled in clinical trial within 3 months of baseline
* Contralateral knee arthritis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
VAS pain scale | 0, 2, 6, 12, 18, 26 weeks

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score | 0, 2, 6, 12, 18, 26 weeks
SF-36® Health Survey | 0, 2, 6, 12, 18, 26 weeks
Physical Examination | 0, 2, 6, 12, 18, 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Grant Jones, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Sports Medicine Center, Columbus, Ohio, United States